CLINICAL TRIAL: NCT01974375
Title: Randomized, Open Label, Non-inferiority Study of Micafungin Versus Fluconazole for the Korean Prevention of Invasive Fungal Disease in Living Donor Liver Transplant Recipients
Brief Title: Micafungin Versus Fluconazole for Prevention of Invasive Fungal Disease in Living Donor Liver Transplant Recipients
Acronym: KOPIN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Giwon Song, Dr., Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MYC-LT-01
Record Dates: First submitted 2013-10-18; First posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Liver Transplant Recipient
Keywords: Living donor; Liver transplant; antifungal prevention
MeSH Terms: interventions — Micafungin; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- micafungin (Experimental): micafungin sodium IV (Mycamine®)
  Interventions: Drug: micafungin
- Fluconazole (Active Comparator): Fluconazole IV (use same brand in each hospital)
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: micafungin — Micafungin 100 mg/day intravenous (2.0 mg/kg/day in subjects weighing <40 kg)
  Other Names: Mycamine
  Arms: micafungin
Drug: Fluconazole — Fluconazole 100~200mg/day, IV care until oral medication becomes possible
  Arms: Fluconazole

SUMMARY:
The purpose of this study is to demonstrate non-inferiority of micafungin at a dose of 100 mg/day versus fluconzeole for the prevention of Invasive Fungal Disease, defined according to the revised EORTC/MSG criteria, undergoing living-donor liver transplantation.

DETAILED DESCRIPTION:
This is Randomized, Open label, Non-inferiority Study of Micafungin versus Fluconazole for the Korean Prevention of Invasive Fungal Disease in Living Donor Liver Transplant Recipients

After transplant subjects will be randomized to one of the following treatment arms:

* Micafungin 100 mg/day intravenous (2.0 mg/kg/day in subjects weighing <40 kg)
* Fluconazole 100~200mg/day, IV care until oral medication becomes possible

Stratification according to centers. Antifungal prophylaxis will be administered once daily for a period of 21 days, or until hospital discharge, whichever occurs first.

This is an open label study; Study center personnel will not be blinded to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years.
* Undergoing Living Donor Liver Transplantation(LDLT)

Exclusion Criteria:

* Any systemic antifungal therapy (excluding fluconazole or SDD for a maximum of 7 days) within 14 days prior to randomization.
* Evidence of documented ('proven' or 'probable') or suspected ('possible') IFD (according to the EORTC/MSG criteria).
* Allergy, hypersensitivity, or any serious reaction to an echinocandin antifungal, or any of the study drugs or their excipients.
* Reimplantation or orthotopic transplantation patient.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Prevention of invasive fungal disease | 6 months
  To demonstrate non-inferiority of micafungin at a dose of 100 mg/day versus fluconzeole for the prevention of Invasive Fungal Disease, defined according to the revised EORTC/MSG criteria, undergoing living-donor liver transplantation.
  'Clinical success' at the End of Prophylaxis as assessed by the investigator.
  Absence of a 'proven' or 'probable' IFD AND No initiation of antifungal treatment (additional antifungal medication or increase in the dose of the study drug due to lack of efficacy)

SECONDARY OUTCOMES:
no events of proven/probable IFD | 6 months
  no events of proven/probable IFD at end of prophylaxis visit and end of study visit
ime to proven/probable IFD | 6 months
  Time to proven/probable IFD
fungal-free survival | 6 months
  fungal-free survival et end of study/and long-term follow-up visit
incidence of superficial mycosis infection and colonization | 6 months
  incidence of superficial mycosis infection and colonization at the end of prophylaxis compare to baseline
saftey by variables | 6 months
  saftey by variables of viatl sign/physical examination/laboratory test
cases of adverse events | 6 months
  cases of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: SUNG-GYU LEE, Professor, Principal Investigator — Asan Medical Center; Giwon Song, Professor, Principal Investigator — Asan Medical Center; Namjoon Lee, Professor, Principal Investigator — Seoul National University; Jaewon Joh, Professor, Principal Investigator — Samsung Medical Center; Dong-Lak Choi, Professor, Principal Investigator — Daegu Catholic University Medical Center; Myung Soo Kim, professor, Principal Investigator — Severance Hospital
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kang WH, Song GW, Lee SG, Suh KS, Lee KW, Yi NJ, Joh JW, Kwon CHD, Kim JM, Choi DL, Kim JD, Kim MS. A Multicenter, Randomized, Open-Label Study to Compare Micafungin with Fluconazole in the Prophylaxis of Invasive Fungal Infections in Living-Donor Liver Transplant Recipients. J Gastrointest Surg. 2020 Apr;24(4):832-840. doi: 10.1007/s11605-019-04241-w. Epub 2019 May 7. PMID 31066013